CLINICAL TRIAL: NCT03492788
Title: Optimizing Cardiac Resynchronization Therapy With Electrocardiographic Imaging
Brief Title: Optimizing CRT With ECGI
Acronym: optCRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study lost access to ECGI
Sponsor: Washington University School of Medicine (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201712146
Record Dates: First submitted 2018-01-17; First posted 2018-04-10 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure, Systolic; Left Bundle-Branch Block
Keywords: cardiac resynchronization therapy; electrocardiographic imaging
MeSH Terms: conditions — Heart Failure, Systolic; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECGI-optimized VV-offset (Active Comparator)
  Interventions: Other: ECGI-optimized VV-offset
- Zero VV-offset (Placebo Comparator)
  Interventions: Other: Zero VV-offset

INTERVENTIONS:
Other: ECGI-optimized VV-offset — ECGI guided optimization of VV offset programming of CRT device
  Arms: ECGI-optimized VV-offset
Other: Zero VV-offset — Standard-of-care nominal (zero VV-offset) programming of CRT device
  Arms: Zero VV-offset

SUMMARY:
CRT is delivered from two electrodes on opposite sides of the heart [right (RV) and left ventricle (LV)] delivering stimulation for more efficient heart beats. There is flexibility in the sequence and temporal staggering of the stimulation from these two electrodes with a different optimum for different patients. However, standard techniques to figure out the optimal stimulation strategy like standard 12-lead surface electrical recording (ECG) or routine ultrasound have failed. The investigators have developed ECG imaging (ECGI) with 250 electrode surface recording combined with CT scan to reconstruct high resolution 4-dimensional panoramic electrical maps of the heart. The study seeks to enroll 56 patients undergoing CRT in a clinical trail to evaluate short and long term impact of using ECGI for optimal programming of CRT.

DETAILED DESCRIPTION:
Heart failure (HF) with reduced ejection fraction is a major global health problem. Every year, over 200,000 patients with HF and electrical abnormalities receive device implants for Cardiac Resynchronization Therapy (CRT). However, one-third of these patients receiving CRT fail to clinically improve, a large population with refractory HF symptoms, high mortality, and tremendous healthcare costs. The overall objective of the study is to improve the clinical response to CRT by physiological optimization of CRT programming with individualized ventriculo-ventricular (VV) offset, guided by novel 4-dimensional panoramic electroanatomical heart mapping using Electrocardiographic Imaging (ECGI). ECGI is a high-resolution, non-invasive, validated technique using 250 recording electrodes combined with heart-torso anatomy from chest CT.

Specific Aims:

1. Assess the acute impact of ECGI-guided CRT optimization on hemodynamic heart function.
2. Determine the impact of ECGI-guided CRT optimization on reverse heart remodeling at 6 months.

Methods:

The study will enroll 56 adult patients undergoing CRT for standard clinical indications.

1. Compare the impact of ECGI-guided CRT optimization vs. standard-of-care (zero VV offset) on acute hemodynamic function i.e. left ventricular stroke volume on Doppler echocardiography.
2. Randomize patients to (a) ECGI-guided CRT optimization or (b) standard-of-care (zero VV offset). Patients will be crossed-over at 6 months and serve as their own controls. The primary outcome will be the difference in heart remodeling, i.e. % reduction of left ventricular end-systolic volume (LVESV) from baseline, between the two groups after 6 months. Reduction in LVESV is a validated physiological marker of CRT response that strongly predicts lower mortality and HF events. The secondary outcomes will include quality-of-life (Kansas City Cardiomyopathy Questionnaire), functional performance (6-minute hall walk distance) and a prognostic biomarker (serum N-terminal proBNP).

The results of this important study will provide key mechanistic insights on the salutary effects of CRT on reverse heart remodeling and enhance the understanding of failure in CRT response. Physiologically tailored CRT therapy would improve individual patient health by reducing CRT non-responders, and decrease the economic burden of refractory HF.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age who are able to give consent, having systolic heart failure despite treatment with guideline directed medical therapy, undergoing successful CRT device implant for standard clinical indications, expected to have over 95% heart beats resynchronized by the pacing device (absence of competing arrhythmias), and have RV or LV pacing latency (stimulus to rapid QRS deflection) ≥30 msec

Exclusion Criteria:

* Patients unable to comply with the study follow-up, life expectancy ≤1 year, suboptimal LV lead location (septal or apical)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
LV reverse remodeling | 6 months
  Echocardiographically evaluated % reduction in LV end-systolic volume (LVESV) from baseline is the primary outcome measure. A reduction in the LVESV is a validated surrogate marker of improved HF outcomes including reduced hospitalizations and increased survival.

SECONDARY OUTCOMES:
Quality-of-life | 6 months
  The validated standardized abbreviated Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) is a secondary outcome measure. The KCCQ-12 is a self-reported disease-specific health status measure for patients with HF. The overall summary KCCQ-12 score ranges from 0 (poor) to 100 (excellent) and represents the summation of the patient's physical limitation, symptom frequency, quality of life and social limitation. Improvement in the KCCQ-12 overall summary score as compared to the baseline will be assessed.
Functional performance | 6 months
  A standard six-minute hall walk distance (meters) will be measured at baseline and at followup to assess increase in walking distance as a reproducible measure of functional performance.
Prognostic biomarker | 6 months
  Serum N-terminal proBNP is a validated prognostic biomarker that is elevated with worsening HF and is associated with worse outcomes including mortality. The NT-proBNP level at followup will be compared to baseline as a marker of improvement in heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Noheria, MBBS, SM, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided